CLINICAL TRIAL: NCT00004801
Title: Phase I/II Study of Monoclonal Factor IX Concentrate for Factor IX Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11956; UNCCH-621
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Hemophilia B; Factor IX Deficiency
Keywords: hematologic disorders; rare disease
MeSH Terms: conditions — Hemophilia B; Hematologic Diseases; Rare Diseases

INTERVENTIONS:
Drug: monoclonal factor IX replacement therapy

SUMMARY:
OBJECTIVES:

Assess the safety and long-term efficacy of monoclonal factor IX concentrate in patients with factor IX deficiency.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive monoclonal factor IX replacement therapy as inpatients. Patients with a satisfactory response receive further therapy as needed for bleeding for up to 36 months at home.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Patients with factor IX deficiency.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3
Dates: Start 1992-03

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert C. White, Study Chair — University of North Carolina